CLINICAL TRIAL: NCT04132817
Title: A Phase 1 Multi-Targeted Study to Promote Anti-Tumor Immunity in ER Positive, HER2 Negative Advanced Breast Cancer
Brief Title: A Study of Multiple Immune and Disease Treatment Combinations in Participants With ER+HER2- Breast Cancer That Has Spread
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA048-001
Record Dates: First submitted 2019-10-02; First posted 2019-10-21 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Nivolumab; Ipilimumab; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A Target class A-1: Nivolumab+nab-paclitaxel (Experimental): The CA048-001 clinical study will utilize a master protocol and subprotocols representing distinct mechanisms of actions. Each subprotocol will contain 1 Group, representing a particular mechanism of action, and will consist of 3 treatment arms that will be simultaneously evaluated. One treatment within a group will be selected to move forward to the next sub-protocol based on safety and tolerability, pharmacodynamic and efficacy data. Thus, the number of treatments within each group is increased by one for each subsequent group, with the intent to simultaneously impact a wide range of mechanisms thought to be important for generating anti-tumor immune responses.
  Interventions: Biological: Nivolumab; Drug: Nab-paclitaxel
- Group A Target Class A-2: Nivolumab+nab-paclitaxel+ipilimumab (Experimental): The CA048-001 clinical study will utilize a master protocol and subprotocols representing distinct mechanisms of actions. Each subprotocol will contain 1 Group, representing a particular mechanism of action, and will consist of 3 treatment arms that will be simultaneously evaluated. One treatment within a group will be selected to move forward to the next sub-protocol based on safety and tolerability, pharmacodynamic and efficacy data. Thus, the number of treatments within each group is increased by one for each subsequent group, with the intent to simultaneously impact a wide range of mechanisms thought to be important for generating anti-tumor immune responses.
  Interventions: Biological: Nivolumab; Biological: Ipilimumab; Drug: Nab-paclitaxel
- Group A Target Class A-3: Nivolumab+nab-paclitaxel+ipilimumab (Experimental): The CA048-001 clinical study will utilize a master protocol and subprotocols representing distinct mechanisms of actions. Each subprotocol will contain 1 Group, representing a particular mechanism of action, and will consist of 3 treatment arms that will be simultaneously evaluated. One treatment within a group will be selected to move forward to the next sub-protocol based on safety and tolerability, pharmacodynamic and efficacy data. Thus, the number of treatments within each group is increased by one for each subsequent group, with the intent to simultaneously impact a wide range of mechanisms thought to be important for generating anti-tumor immune responses.
  Interventions: Biological: Nivolumab; Biological: Ipilimumab; Drug: Nab-paclitaxel

INTERVENTIONS:
Biological: Nivolumab — specified dose on specified days
Biological: Ipilimumab — specified dose on specified days
  Arms: Group A Target Class A-2: Nivolumab+nab-paclitaxel+ipilimumab; Group A Target Class A-3: Nivolumab+nab-paclitaxel+ipilimumab
Drug: Nab-paclitaxel — specified dose on specified days

SUMMARY:
The hypothesis of the CA048-001 Phase 1 clinical trial is targeting multiple mechanisms involved in generating and maintaining antitumor immune response will lead to a tolerable and robust anti-tumor response. This study utilizes an innovative clinical trial design to determine the safety, tolerability, pharmacodynamic activity and efficacy of targeting multiple, distinct combination regimens that modulate several immune and non-immune mechanisms by escalating the number of therapies administered.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histological and cytological confirmation of adenocarcinoma of the breast
* Documented HER2 negative and estrogen receptor (ER) positive status of primary or metastatic tumor tissue using the most recently assessed tumor specimen, according to the local laboratory parameters
* ER negativity is defined as < 1% of tumor cells expressing hormonal receptors via IHC analysis
* At least one measurable lesion, as per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST v1.1] that can be accurately assessed at baseline and is suitable for repeated assessment by computed tomography (CT) or magnetic resonance imaging (MRI)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Women and Men must agree to follow specific methods of contraception, if applicable, while participating in the trial

Exclusion Criteria:

* Allergy or hypersensitivity to any study drugs or their excipients
* Any other sound medical, psychiatric and/or social reason as determined by the investigator
* Active, known, or suspected autoimmune disease or immune-related diseases
* History of unstable or deteriorating cardiac disease within the previous 12 months prior to screening
* Prior therapy with anti-programmed death 1 (PD-1), anti-programmed death-ligand 1 (PD-L1) or anti-Cytotoxic T Lymphocyte Antigen 4 (CTLA-4) class antibody
* Any major surgery within 4 weeks of the first dose of study treatment

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 3 years
Incidence of Serious Adverse Events (SAEs) | Up to 3 years
Incidence of AEs leading to dose and asset limiting toxicity (DALT) | 8 weeks following initial dose
Incidence of AEs leading to discontinuation | Up to 3 years
Incidence of laboratory abnormalities | Up to 3 years

SECONDARY OUTCOMES:
Change from baseline in programmed cell death receptor-ligand 1 (PD-L1) by immunohistochemistry (IHC) | Day 0, Day 22, Day 50
Objective Response Rate (ORR) | 24 weeks
Median duration of response (mDOR) | 24 weeks
Progression-free survival rate (PFSR) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- United States (8):
  - Local Institution, Los Angeles, California
  - Local Institution - 0003, Sacramento, California
  - Local Institution - 0009, Aurora, Colorado
  - Local Institution - 0002, St Louis, Missouri
  - Local Institution - 0008, New York, New York
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Dallas, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm